CLINICAL TRIAL: NCT02136407
Title: Seasonal Variations in Serum 25-hydroxy Vitamin-D Levels in a Swedish Cohort
Status: Completed | Type: Observational
Sponsor: Sahlgrenska University Hospital (Other)
Responsible Party: Principal Investigator, Eva Klingberg, MD, PhD, Sahlgrenska University Hospital
Other Study IDs: EPN399-09
Record Dates: First submitted 2014-05-02; First posted 2014-05-13 (Estimated); Last update posted 2014-05-13 (Estimated); Status verified 2014-05

CONDITIONS: Vitamin-D Insufficiency
Keywords: Vitamin D; vitamin D deficiency; parathyroid hormone
MeSH Terms: conditions — Vitamin D Deficiency

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — Serum
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Blood donors: N=540
- Thrombocyte donors: N=75

SUMMARY:
The purpose of this study was to study seasonal inter-individual and intra-individual variations in S-25(OH)D and to explore parameters associated with S-25-OHD in healthy Swedish adults.

DETAILED DESCRIPTION:
Serum was collected during 12 months and analysed for 25(OH)D in 540 healthy blood donors. The blood donors answered questionnaires concerning vitamin D supplements, smoking, physical activity, sunbed use and holidays in sunny locations. Repeated serum samples were also collected from thrombocyte donors to study the intra-individual variations in S-25(OH)D.

ELIGIBILITY:
Inclusion Criteria:

* healthy at the time of donating blood

Exclusion Criteria:

* unhealthy

Ages: 16 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Blood donors
Sampling Method: Probability Sample
Enrollment: 615 (Actual)
Dates: Start 2009-10; Primary Completion 2010-09 (Actual); Study Completion 2010-09 (Actual)

PRIMARY OUTCOMES:
Inter-individual and intra-individual varations in serum 25-hydroxy vitamin-D during different seasons. | Group1:Blood donors, single test, 25(OH)vit D at inclusion . Group 2: thrombocyte donors: multiple tests, serum 25(OH)vit D during 8 months.

CONTACTS AND LOCATIONS:
Locations (1):
- Sahlgrenska University Hospital, Gothenburg, Sweden